CLINICAL TRIAL: NCT01059942
Title: Development and Validation of a Tool to Evaluate Hand-off Quality
Brief Title: Development and Validation of a Tool to Measure Hand-off Quality
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 09-258-A; 1R03H5018278-01 (Other Grant/Funding Number: The Agency for Healthcare Research and Quality)
Record Dates: First submitted 2010-01-27; First posted 2010-02-01 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Communication; Patient Care; Quality of Health Care
Keywords: communication barriers; clinical competence; medical education; internship and residency; hospitalist; Quality Assurance, Healthcare; Patient Care; Internal Medicine
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalist physicians/house-staff: Consented Academic Hospitalist and Internal Medicine Residency staff
  Interventions: Other: mock handoff exposure; Other: Introduction of CEX tool in Actual Hand-offs

INTERVENTIONS:
Other: mock handoff exposure — Attending and house-staff physicians will analyze six video scenarios using the Hand-off CEX, rating each of the dimensions of hand-off competence for both the senders and receivers of the mock hand-off.
Other: Introduction of CEX tool in Actual Hand-offs — We will teach hospitalist physicians and house-staff how to utilize the Hand-off CEX in conducting their own hand-offs.

SUMMARY:
The aim of this project is to develop and validate a simple, flexible, reliable, real-time observation tool to evaluate hand-off practices. The Hand-off CEX is a paper-based instrument that can be used to evaluate either the sender or the receiver of hand-off communication. This tool is based on a previously-validated, widely-used, real-time educational evaluation tool (the Mini-CEX); published expert opinion; and our prior research . The investigators' tool incorporates unique role-based anchors for both senders and receivers that refer to verbal communication, professionalism and environment, hand-off domains informed by preliminary work and expert opinion. The Hand-off CEX(Clinical Evaluation Exercise) will be used by academic hospitalists and house-staff physicians to assess feasibility. We, the investigators, will also assess the construct validity and inter-rater reliability of the tool through the use of standardized, videotaped hand-off scenarios depicting various levels of performance of a hand-off scenario.

We hypothesize that the Hand-off CEX will arm educators with an innovative, necessary, valid and feasible method for training health professionals to conduct safe and effective hand-offs. Finally, the Hand-off CEX will be a useful tool to assist hospitals in improving patient safety.

DETAILED DESCRIPTION:
Transitions of patient care among inpatient providers occur frequently and require providers to transmit critical clinical information. If information is omitted or misunderstood during a hand-off, serious clinical consequences may result for patient care. In fact, studies have shown that hand-offs are often variable and represent a major gap in safe patient care. For patients cared for by resident physicians, dangers posed by poor communication may be amplified since the implementation of resident duty hour restrictions in July 2003 has increased transfer frequency.In addition, few trainees receive formal training on hand-offs. The Joint Commission currently requires hospitals to implement a standardized, interactive approach to hand-off communications. Unfortunately, due to a lack of valid, standardized tools to evaluate hand-off quality, hospitals and educators cannot assess whether their hand-offs meet these criteria. More recently, the Institute of Medicine has recommended that all residents receive formal education on hand-off strategies.

Education about best practices during hand-offs and assessment of hand-off quality is needed for several reasons: to improve clinical practice through evaluation and feedback, to illuminate areas of deficiency in current practices and to maximize patient safety in this era of duty hour restrictions. At the University of Chicago and Yale, investigators have extensive experience in describing hand-off quality, designing and implementing novel curricula to improve hand-off education amongst varying levels of trainees and have elucidated the relationship between patient care outcomes and poor hand-off quality. Therefore, drawing from our preliminary work in this area, and relevant practices in other industries, we aim to develop and test a generalizable tool to evaluate hand-offs in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* All academic hospitalist and internal medicine house-staff are eligible to participate.

Exclusion Criteria:

* We have no exclusion criteria. All internal medicine residents and hospitalist physicians at the University of Chicago will be invited to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Academic Hosptialists and Internal Medicine Residents of the University of Chicago Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Residents and Hospitalists will use the Hand-off CEX to conduct evaluations of their sign-out process. In addition, each hand-off will be evaluated simultaneously by a trained observer. | January 2010-January 2015

SECONDARY OUTCOMES:
Upon completion of the Hand-Off evaluation, participants and observers will be asked about their overall satisfaction with the evaluation. This will be a marker of the feasibility of the Hand-Off CEX. | January 2010-January 2015
For the validity part of the study, attending and house-staff physicians will analyze six video scenarios using the Hand-off CEX, rating each of the dimensions of hand-off competence for both the senders and receivers of the handoff. | January 2010-January 2015

CONTACTS AND LOCATIONS:
Overall Officials: Vineet M Arora, MD, MA, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States